CLINICAL TRIAL: NCT02010177
Title: Clinical Outcome of Patients With Low Ejection Fraction or Low-gradient Severe Aortic Stenosis
Brief Title: Clinical Outcome of Patients With Low-gradient Severe Aortic Stenosis
Status: Suspended | Type: Observational
Why Stopped: No recruitment
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-13-0686-IB-CTIL
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-06

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the ability of baseline clinical parameters and imaging modalities to predict short and long term left ventricular function and clinical outcome of subjects with low-gradient, severe aortic stenosis.

To assess the impact of aortic valve replacement as compared to medical therapy on clinical outcome of patients with low-gradient, severe aortic stenosis.

To assess possible impact of aortic annulus assessment using 3-dimensional imaging modalities on the assessment of AS severity and definition of low gradient severe aortic stenosis.

DETAILED DESCRIPTION:
To assess the ability of baseline clinical parameters and imaging modalities to predict short and long term left ventricular function and clinical outcome of subjects with impaired left ventricular function and / or low-gradient, severe aortic stenosis.

To assess the impact of aortic valve replacement as compared to medical therapy on clinical outcome of patients with impaired left ventricular function and / or low-gradient, severe aortic stenosis.

To assess possible impact of aortic annulus assessment using 3-dimensional imaging modalities on the assessment of AS severity and definition of low gradient severe aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis defined as aortic valve area of less than 1 cm2 or index area of 0.6 cm2/m2 and low gradient (mean gradient across the aortic valve <40 mmHg) by echocardiography
2. Symptomatic patients with aortic stenosis referred for medically indicated AVR
3. Signed informed consent to participate in the study.

Exclusion Criteria:

1. Pregnancy or breast feeding (women of childbearing potential will have a serum or urine pregnancy test).
2. Need for emergency surgery for any reason.
3. Any case in which the practicing physician asserts that enrollment in the protocol will adversely affect the patient treatment course.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with severe symptomatic aortic stenosis defined as aortic valve area of less than 1 cm2 or index area of 0.6 cm2/m2 by echocardiography, together with low-gradient (mean gradient across the aortic valve <40 mmHg) who are referred for treatment of AS will be recruited. A total of up to 100 consecutive subjects of both genders will be enrolled at the Sheba Medical Center. The study procedures, clinical management and follow up will be done at the Sheba Medical Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2022-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction after aortic valve replacement | 2±1 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel